CLINICAL TRIAL: NCT02431299
Title: Illness Management and Recovery Treatment Integrity Scale Validation and Leadership Intervention Development
Acronym: IT IS VALID
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Alan McGuire, Research Scientist, Indiana University
Other Study IDs: 1R21MH096835-01 (NIH)
Record Dates: First submitted 2015-04-23; First posted 2015-05-01 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-11

CONDITIONS: Severe Mental Illness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Illness Management and Recovery (IMR) is an evidenced-based approach to teaching consumers with severe mental illness how to set and achieve personal recovery goals and acquire the knowledge and skills to independently manage their illnesses. Longitudinal, multi-site, and randomized controlled trials have shown IMR to be effective in increasing illness self-management and coping; some evidence also points to reduced hospitalization rates. Fidelity, or adherence to a specific treatment model, is equally important to both clinical research and to the practical dissemination of evidence-based practices to the field.

To this end, the research team has developed an IMR clinician-level fidelity assessment, the IMR Treatment Integrity Scale (IT-IS). However, the validity of the preliminary IT-IS has not been rigorously evaluated. Additionally, it is crucial to develop strategies to utilize the IT IS to increase adherence to the IMR model and ultimately increase consumer outcomes.

The purpose of this study is to assess the construct validity of the IT-IS by testing the relationship between IT-IS elements and mechanisms of change and proximal outcomes. The investigators will collect a sample of IMR session recordings and pre-post data from IMR participants from recruitment sites in Indiana, New Jersey and several other states. The investigators will test hypothesized relationships between specific program elements and theoretically proposed mechanisms of change. The investigators will also assess organizational and clinician factors affecting IMR competence by including a survey for the staff members who are located as sites where the investigators have clinicians participating in providing IMR.

ELIGIBILITY:
Inclusion Criteria:

Clinicians:

* 18 years or older
* Providing IMR individually or in group format at a participating agency
* Willing and able to provide consent
* Willing to complete study measures
* Willing to be audio recorded

Consumers:

* 18 years or older
* Willing and able to provide consent
* Able to complete a brief cognitive screener
* Willing to complete study measures
* Receiving IMR intervention at a participating agency
* Willing to be audio recorded

Exclusion Criteria:

* Individuals younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consumers with mental illness, who are participating in the Illness Management and Recovery intervention in New Jersey and Indiana. This includes consumers from state hospitals, rehabilitation centers and community mental health centers. Additionally, the clinicians who are leading the intervention are considered to be participants of the study as well.
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- IMR Consumers: Consumer participants who are engaging in Illness Management and Recovery (IMR) intervention.
- IMR Clinicians: The clinicians who provided IMR intervention to the IMR Consumers
Period: Overall Study
Arm/Group | IMR Consumers | IMR Clinicians
Started | 236 | 63
Completed | 183 | 62
Not Completed | 53 | 1

BASELINE CHARACTERISTICS:
Population: One clinician did not complete the baseline measures, thus leaving us the baseline characteristics for 62 IMR Clinicians. The only baseline measure collected for the IMR Clinicians were demographic variables (i.e. Age, Gender, Region of Employment). The remaining outcome measures aren't collected because they are specific to the patient population.
Groups:
- IMR Clinicians: Clinicians who provided the IMR intervention to the IMR Consumers
- Total: Total of all reporting groups
Arm/Group | IMR Consumers | IMR Clinicians | Total
Number analyzed (Participants) | 236 | 62 | 298
Age, Categorical [Count of Participants; unit: Participants] — Every attempt was made to collect this information from all participants, however this data was missing in some instances. Data was collected via self-report, and thus if the question was omitted by the participant the data was not available for analyses.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 231 | 61 | 292
    >=65 years | 5 | 1 | 6
Gender [Number; unit: participants] — Every attempt was made to collect this information from all participants, however this data was missing in some instances. Data was collected via self-report, and thus if the question was omitted by the participant the data was not available for analyses.
  participants
    Female | 90 | 41 | 131
    Male | 128 | 21 | 149
Region of Enrollment [Number; unit: participants] — Every attempt was made to collect this information from all participants, however this data was missing in some instances. Data was collected via self-report, and thus if the question was omitted by the participant the data was not available for analyses.
  participants
    United States | 236 | 62 | 298
Illness Management and Recovery Scale [Mean (Standard Deviation); unit: units on a scale] — This measure is designed to assess consumer-rated illness self management skills. This scale is based on a 15 items, each rated on a 5 point Likert scale, ranging from 1 to 5. Higher numbers of this scale represent better outcomes. A mean score of all 15 items is provided as the primary outcome score for this scale.
  units on a scale | 3.55 (.6) | NA (NA) — Data not collected for clinicians | 3.55 (.6)
Working Alliance Inventory Short Form [Mean (Standard Deviation); unit: units on a scale] — This is a consumer rated scale indicated working alliance between consumer and clinician. The scale has 12 items, rated on a 7 point Likert style scale (ranging from 1-7). The total score provided a mean score of all 12 items. Better working alliance is indicated by a higher score.
  units on a scale | 5.65 (1.0) | NA (NA) — Data not collected for clinicians | 5.65 (1.0)
Multidimensional Scale of Perceived Social Support [Mean (Standard Deviation); unit: units on a scale] — This scale is a consumer rated assessment of perceived social support systems. There are 12 items each rated on a 7 point Likert scale (ranging from 1-7). A mean score is calculated from all 12 items. Higher scores represent better outcomes (i.e. higher levels of perceived social support).
  units on a scale | 4.94 (1.7) | NA (NA) — Data not collected for clinicians | 4.94 (1.7)
Adult State Hope Scale [Mean (Standard Deviation); unit: units on a scale] — This is a consumer rated measure that assesses the level of goal related hope a consumer possesses. This version is a 6 item measure, with each item rated on a 4 point scale (range 1-4, with 1 being "Definitely False" and 4 being "Definitely True"). A summary score is calculated by summing all 6 items. Higher scores represent better outcomes (i.e. higher goal related hope). These summary scores were then averages to calculate a mean score for our sample.
  units on a scale | 18.8 (3.7) | NA (NA) — Data not collected for clinicians | 18.8 (3.7)
Medication Adherence Rating Scale [Mean (Standard Deviation); unit: units on a scale] — This is a consumer rated scale assessing medication adherence. This is a 10 item scale with each question rated as "yes" or "no". A yes is assigned a value of 1. The scale ranges from 0 (no "yes" responses) to 10 (all "yes" responses endorsed). The total number of "yes" responses is totaled to create a summary score. The mean score is calculated based on averaging the summary scores for the entire consumer sample. Higher scores mean better outcomes for medication adherence.
  units on a scale | 2.45 (.12) | NA (NA) — Data not collected for clinicians | 2.45 (.12)
UNCOPE [Mean (Standard Deviation); unit: units on a scale] — This measure is a consumer rated substance abuse screener consisting of 6 "yes" or "no" questions. A response of "yes" is assigned a value of 1. The total number of "yes" responses are summed and a score of greater than 4 indicates likelihood of substance abuse. Higher scores mean worse outcomes for this scale (i.e. the higher the score, the greater the likelihood of substance abuse issues).
  units on a scale | 1.88 (.13) | NA (NA) — Data not collected for clinicians | 1.88 (.13)
Brief COPE Inventory Adaptive Coping Subscale [Mean (Standard Deviation); unit: units on a scale] — This is a consumer rated assessment of adaptive coping skills. This is derived from the 28 item, full scale. The scale uses a 1-4 Likert scale, indicating the frequency of using different coping strategies. There are 14 subscales, each calculated by summing 2 items. The range on each subscale is 2 - 8. The 14 subscales are further combined into 2 larger scales - maladaptive and adaptive coping. Adaptive coping is calculated by averaging the responses from 8 out of the 14 subscales. Higher scores indicate better outcomes (i.e. higher use of adaptive coping strategies).
  units on a scale | 5.64 (1.4) | NA (NA) — Data not collected for clinicians | 5.64 (1.4)
Brief COPE Inventory Maladaptive Coping Subscale [Mean (Standard Deviation); unit: units on a scale] — This is a consumer rated assessment of adaptive coping skills. This is derived from the 28 item, full scale. The scale uses a 1-4 Likert scale, indicating the frequency of using different coping strategies. There are 14 subscales, each calculated by summing 2 items. The range on each subscale is 2 - 8. The 14 subscales are further combined into 2 larger scales - maladaptive and adaptive coping. Maladaptive coping is calculated by averaging the responses from 6 out of the 14 subscales. Higher scores indicate worse outcomes (i.e. higher use of maladaptive coping strategies).
  units on a scale | 4.46 (1.2) | NA (NA) — Data not collected for clinicians | 4.46 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Illness Management and Recovery Scale
Description: Post-intervention scores were assessed. This measure is designed to assess consumer-rated illness self management skills. This scale is based on a 15 items, each rated on a 5 point Likert scale, ranging from 1 to 5. Higher numbers of this scale represent better outcomes. A mean score of all 15 items is provided as the primary outcome score for this scale.
Time Frame: 3-Months
Population: Every effort was made to collect post-intervention follow up data for participants. In some instances, participants were unable to provide this information (i.e. hospitalized, unable to attend data collection session, unwilling). As all outcome measures were consumer self-rated, if the consumer was unavailable data is missing for that participant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IMR Consumers
Number analyzed (Participants) | 183
units on a scale | 3.72 (0.5)
Statistical Analysis 1: Comparison: IMR Consumers; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — Whether there were significant changes in the IMRS baseline scores to IMRS follow up scores; t = 2.78, df = 182

2. Primary Outcome: Illness Management and Recovery Treatment Integrity Scale
Description: Clinician competency rating scale was used to assess clinician competence in providing IMR. This data was used to test the theory that IMR competency would impact consumers' ability to engage in illness self management practices as rated by the Illness Management and Recovery Scale. This scale is rated by trained observers, and the scale contains 16 items, rated on a 1 - 5 point scale. A 5 indicates higher competency and fidelity to the IMR treatment model. A mean score is calculated across all 16 items. Higher scores indicate higher clinician competence in providing IMR.
Time Frame: 3-Months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- IMR Clinicians: Clinicians providing IMR to the IMR consumers.
Arm/Group | IMR Clinicians
Number analyzed (Participants) | 63
units on a scale | 2.73 (.55)
Statistical Analysis 1: Comparison: IMR Clinicians; Hypothesized that higher levels of IMR competence would predict higher IMRS outcomes; Test type: Superiority or Other; p < 0.05, Regression, Linear

3. Secondary Outcome: Working Alliance Inventory Short Form
Description: This is a consumer rated scale indicated working alliance between consumer and clinician. The scale has 12 items, rated on a 7 point Likert style scale (ranging from 1-7). The total score provided a mean score of all 12 items. Better working alliance is indicated by a higher score.
Time Frame: 3-Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IMR Consumers
Number analyzed (Participants) | 158
units on a scale | 5.58 (1.0)

4. Secondary Outcome: Multidimensional Scale of Perceived Social Support
Description: This scale is a consumer rated assessment of perceived social support systems. There are 12 items each rated on a 7 point Likert scale (ranging from 1-7). A mean score is calculated from all 12 items. Higher scores represent better outcomes (i.e. higher levels of perceived social support).
Time Frame: 3-Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IMR Consumers
Number analyzed (Participants) | 183
units on a scale | 5.18 (.11)

5. Secondary Outcome: Adult State Hope Scale
Description: This is a consumer rated measure that assesses the level of goal related hope a consumer possesses. This version is a 6 item measure, with each item rated on a 4 point scale (range 1-4, with 1 being "Definitely False" and 4 being "Definitely True"). A summary score is calculated by summing all 6 items. Higher scores represent better outcomes (i.e. higher goal related hope). These summary scores were then averages to calculate a mean score for our sample.
Time Frame: 3-Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IMR Consumers
Number analyzed (Participants) | 181
units on a scale | 19.13 (3.6)

6. Secondary Outcome: Brief COPE Adaptive Subscale
Description: This is a consumer rated assessment of adaptive coping skills. This is derived from the 28 item, full scale. The scale uses a 1-4 Likert scale, indicating the frequency of using different coping strategies. There are 14 subscales, each calculated by summing 2 items. The range on each subscale is 2 - 8. The 14 subscales are further combined into 2 larger scales - maladaptive and adaptive coping. Adaptive coping is calculated by averaging the responses from 8 out of the 14 subscales. Higher scores indicate better outcomes (i.e. higher use of adaptive coping strategies).
Time Frame: 3-Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IMR Consumers
Number analyzed (Participants) | 183
units on a scale | 5.73 (1.3)

7. Secondary Outcome: Medication Adherence Rating Scale
Description: This is a consumer rated scale assessing medication adherence. This is a 10 item scale with each question rated as "yes" or "no". A yes is assigned a value of 1. The scale ranges from 0 (no "yes" responses) to 10 (all "yes" responses endorsed). The total number of "yes" responses is totaled to create a summary score. The mean score is calculated based on averaging the summary scores for the entire consumer sample. Higher scores mean better outcomes for medication adherence.
Time Frame: 3-Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IMR Consumers
Number analyzed (Participants) | 180
units on a scale | 2.45 (.15)

8. Secondary Outcome: UNCOPE Measure
Description: This meThis measure is a consumer rated substance abuse screener consisting of 6 "yes" or "no" questions. A response of "yes" is assigned a value of 1. The total number of "yes" responses are summed and a score of greater than 4 indicates likelihood of substance abuse. Higher scores mean worse outcomes for this scale (i.e. the higher the score, the greater the likelihood of substance abuse issues).
Time Frame: 3-Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IMR Consumers
Number analyzed (Participants) | 174
units on a scale | .30 (.03)

9. Secondary Outcome: Brief COPE Maladaptive Subscale
Description: This is a consumer rated assessment of adaptive coping skills. This is derived from the 28 item, full scale. The scale uses a 1-4 Likert scale, indicating the frequency of using different coping strategies. There are 14 subscales, each calculated by summing 2 items. The range on each subscale is 2 - 8. The 14 subscales are further combined into 2 larger scales - maladaptive and adaptive coping. Maladaptive coping is calculated by averaging the responses from 6 out of the 14 subscales. Higher scores indicate worse outcomes (i.e. higher use of maladaptive coping strategies).
Time Frame: 3-Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IMR Consumers
Number analyzed (Participants) | 183
units on a scale | 4.47 (1.1)

ADVERSE EVENTS:
Time Frame: Data was collected for 3-months during the study intervention period.
Groups:
- IMR Clinicians: Clinician participants who are providing Illness Management and Recovery (IMR) intervention.
Arm/Group | IMR Consumers | IMR Clinicians
Serious Adverse Events (participants affected / at risk) | 0/236 | 0/63
Other Adverse Events (participants affected / at risk) | 0/236 | 0/63

LIMITATIONS AND CAVEATS:
Unable to randomly assign a level of competency in providing IMR. Geographically limited to three states within the United States. Relatively brief observation period (3-months).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No